CLINICAL TRIAL: NCT01805141
Title: Phase I Pilot Study to Evaluate the Prognostic Value of Perfusion CT for Primary Cervical Cancer
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Other Study IDs: GYNCVX0003; 25821 (Other: Stanford IRB)
Record Dates: First submitted 2013-02-27; First posted 2013-03-06 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Cervical Cancer
Keywords: Cervix Uteri
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The investigators hope to learn whether perfusion CT is a useful way to assess primary cervical tumor microenvironment and whether there is a relationship between pretreatment perfusion CT measurements and primary cervical tumor size, lymph node involvement (as assessed by standard of care pretreatment fludeoxyglucose Positron emission tomography/CT (FDG-PET/CT)), and treatment response (as assessed by standard of care 3-month post-therapy FDG-PET/CT).

ELIGIBILITY:
Inclusion criteria:

* >18 years old
* with biopsy-proven squamous, adenocarcinoma or adenosquamous cervical cancer
* no history of prior pelvic radiation and should be able to receive chemoradiation
* non-pregnant women who have not previously undergone a hysterectomy, as that would have removed the cervix.
* able to give informed consent

Exclusion criteria:

* Subjects whose tumors are not FDG avid on the pre-therapy PET.
* Allergy or inability to receive iodinated CT contrast

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Approximately 12-15 cervical cancer patients are referred for radiation each year.
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2013-08; Primary Completion 2018-10-04 (Actual); Study Completion 2018-10-04 (Actual)

PRIMARY OUTCOMES:
Measure perfusion in primary cervical tumors using perfusion CT. | 3-6 months
  Treatment response will be assessed using a post-treatment FDG-PET/CT to evaluate for complete response, persistent disease or new disease. The association between pre-treatment perfusion CT parameters and response on the post-treatment FDG-PET/CT will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Kidd, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

REFERENCES:
- [Derived] Capaldi DPI, Hristov DH, Kidd EA. Parametric Response Mapping of Coregistered Positron Emission Tomography and Dynamic Contrast Enhanced Computed Tomography to Identify Radioresistant Subvolumes in Locally Advanced Cervical Cancer. Int J Radiat Oncol Biol Phys. 2020 Jul 15;107(4):756-765. doi: 10.1016/j.ijrobp.2020.03.023. Epub 2020 Apr 3. PMID 32251757